CLINICAL TRIAL: NCT01057342
Title: Carboplatin and Paclitaxel Plus ASA404 as First Line Chemotherapy for Extensive-Stage Small-Cell Lung Cancer (ES-SCLC): A Phase II Trial
Brief Title: Paclitaxel, Carboplatin, and Dimethylxanthenone Acetic Acid in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 15/08; SWS-SAKK-15-08; EUDRACT-2009-016960-34; EU-21001; NOVARTIS-CASA404ACCH01T
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Paclitaxel; vadimezan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel, Carboplatin, ASA404 (Experimental)
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: vadimezan

INTERVENTIONS:
Drug: carboplatin — AUC 6 i.v. given after paclitaxel as the second treatment on day 1 of each 3-week cycle.
  Other Names: Paraplatin
Drug: paclitaxel — 175 mg/m2 i.v. first treatment on day 1 of each 3-week cycle.
  Other Names: Abraxane Taxol
Drug: vadimezan — 1800 mg/m2 i.v. following the administration of paclitaxel and carboplatin on day 1 of each 3-week cycle
  Other Names: ASA404

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Dimethylxanthenone acetic acid may stop the growth of small cell lung cancer by blocking blood flow to the tumor. Giving paclitaxel and carboplatin together with dimethylxanthenone acetic acid may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects of giving paclitaxel and carboplatin together with dimethylxanthenone acetic acid and to see how well they work in treating patients with extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the 24-week (6 months) progression-free survival of patients with extensive stage small cell lung cancer treated with paclitaxel, carboplatin, and dimethylxanthenone acetic acid.

Secondary

* To assess efficacy and safety of this regimen in these patients.
* To evaluate predictive molecular markers for gene expression analyses, serum proteomics, and pharmacogenomics. (exploratory)

OUTLINE: This is a multicenter study.

Patients receive paclitaxel IV over 3 hours, carboplatin IV over 30 minutes, and dimethylxanthenone acetic acid IV over 20 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Blood and tissue samples may be collected periodically for predictive molecular markers for gene expression analysis, plasma proteomics, and pharmacogenomics.

After completion of study treatment, patients are followed every 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically (preferred) or cytologically confirmed small-cell lung carcinoma (SCLC) by surgical biopsy, brushing, washing, OR core needle aspiration (sputum cytology alone not acceptable)

  * Extensive stage or stage IV disease, including patients with malignant pleural or pericardial effusion

    * No pleural effusion that causes ≥ CTC grade 2 dyspnea
* Not suitable for potentially curative combined-modality treatment for this disease
* Measurable or non-measurable disease
* No CNS metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Hemoglobin ≥ 10.0 g/dL
* Absolute neutrophils ≥ 2.0 x 10^9/L (without the use of growth factors)
* Platelet count ≥ 100 x 10^9/L
* Bilirubin ≤ 1.5 x the upper limit of normal (ULN)
* ALT ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases)
* Alkaline phosphatase ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases)
* Creatinine clearance ≥ 45 mL/min
* INR ≤ 1.5
* Magnesium, potassium, and calcium (corrected for albumin) normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study therapy
* No recent hemoptysis associated with SCLC (> 1 teaspoon in a single episode within 4 weeks)
* No other malignancy within the past 5 years except for nonmelanoma skin cancer or cervical cancer in situ
* Must not have a history of any of the following conditions:

  * Myocardial infarction within the past 12 months
  * Uncontrolled hypertension (systolic BP > 160 mm Hg and/or diastolic BP > 90 mm Hg) or poor compliance with anti-hypertensive regimen
  * Sustained ventricular tachycardia
  * Ventricular fibrillation or Torsades de Pointes
  * Long QT syndrome
  * QTc of > 450 msec
  * NYHA class III or IV congestive heart failure
  * Unstable or poorly controlled angina pectoris, including Prinzmetal variant angina pectoris
  * Right bundle branch block and left anterior hemiblock (bifascicular block)
  * Bradycardia (defined as heart rate < 50 beats per minute)
  * Cardiac arrhythmias (i.e., symptomatic, but may not require medications) CTCAE grade ≥ 2
* No significant neurologic or psychiatric disorder that would compromise study participation
* No peripheral sensory neuropathy with functional impairment ≥ CTC grade 2 (regardless of cause)
* No concurrent severe and/or uncontrolled medical disease, including any of the following:

  * Uncontrolled diabetes
  * Chronic renal disease
  * Chronic liver disease
  * Confirmed diagnosis of HIV infection
  * Active uncontrolled infection
* No serious underlying medical condition, in the judgment of the investigator, that would impair the patient's ability to participate in the trial
* No known hypersensitivity to study drugs or to any other component of the study drugs (taxanes or other drugs formulated in Cremophor EL [polyoxyethylated castor oil])

PRIOR CONCURRENT THERAPY:

* Recovered from all prior therapy
* No prior systemic chemotherapy, immunotherapy, or biologic anti-cancer therapy
* More than 2 weeks since prior and no concurrent radiotherapy

  * Localized palliative radiotherapy to symptomatic bone metastases allowed
* More than 2 weeks since minor surgery

  * Insertion of a vascular access device allowed
* More than 3 weeks since prior dimethylxanthenone acetic acid for prophylactic cranial irradiation
* More than 4 weeks since major surgery (defined by the use of general anesthesia)
* At least 30 days since prior and no other concurrent investigational drugs or anti-cancer therapy
* No treatment in a clinical trial within 30 days prior to trial entry
* No concurrent therapy with a risk of causing Torsades de Pointes
* No concurrent drugs that would be contraindicated for use with study drugs
* No factors with the potential to prolong QT interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate | at 24 weeks (6 months)
  The status of progression free survival at 24 weeks (+/- 2 weeks) from trial registration will be assessed. A PFS event is defined as (whichever occurs first):
  * Relapse or progression assessed according to the RECIST 1.1 criteria (Appendix 1)
  * Death of any cause.

SECONDARY OUTCOMES:
Adverse events by NCI CTCAE v3.0 | until 30 days after trial therapy end
Best objective response OR complete or partial response according to RECIST 1.1 | whilst receiving the trial therapy
Time to progression | Defined as the time from registration until documented Small-cell Lung Cancer (SCLC) progression or death as a result of SCLC.
Overall survival | Time from registration until death as a result of any cause.
One-year survival rate | at 1 year
  Patients alive one year after trial registration

CONTACTS AND LOCATIONS:
Overall Officials: Martin Frueh, MD, Study Chair — Cantonal Hospital of St. Gallen; Miklos Pless, MD, Study Chair — Kantonsspital Winterthur KSW; Oliver Gautschi, MD, Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (12):
- Switzerland (12):
  - Saint Claraspital AG, Basel
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni, Bellinzona
  - Inselspital Bern, Bern
  - Spitalzentrum Biel, Biel
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Olten, Olten
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Onkologie Schaffhausen, Schaffhausen
  - Regionalspital, Thun
  - Kantonsspital Winterthur, Winterthur
  - Klinik Hirslanden, Zurich

REFERENCES:
- [Result] Fruh M, Cathomas R, Siano M, Tscherry G, Zippelius A, Mamot C, Erdmann A, Krasniqi F, Rauch D, Simcock M, Kuttel E, Fustier P, Pless M; Swiss Group for Clinical Cancer Research. Carboplatin and paclitaxel plus ASA404 as first-line chemotherapy for extensive-stage small-cell lung cancer: a multicenter single arm phase II trial (SAKK 15/08). Clin Lung Cancer. 2013 Jan;14(1):34-9. doi: 10.1016/j.cllc.2012.04.001. Epub 2012 May 24. PMID 22633220